CLINICAL TRIAL: NCT02062996
Title: The Hemodynamic and Pharmacokinetic Analysis of Oxymetazoline Absorption During Functional Endoscopic or Turbinate Reduction Surgery and From the Nasal Mucosa During Operative Dentistry
Brief Title: Hemodynamic and Pharmacokinetic Analysis of Oxymetazoline Absorption
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not receive FDA approval for IND
Sponsor: Richard Cartabuke (Other)
Responsible Party: Sponsor-Investigator, Richard Cartabuke, Co-Director Outpatient Anesthesia Services, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-00016
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Dental Anesthesia; Nasal Surgical Procedures; Intranasal Drug Administration
MeSH Terms: interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- ENT - full strength (Experimental): Full strength oxymetazoline pledgets packed in the nose (total volume 20 ml).
  Interventions: Drug: Oxymetazoline
- ENT - 1/2 strength (Experimental): ½ strength oxymetazoline pledgets packed in the nose (total volume 20 ml).
  Interventions: Drug: Oxymetazoline
- DENTAL - Full strength 1.0 mL (Experimental): Full strength oxymetazoline 1.0 mL to each naris (total =1000 mcg).
  Interventions: Drug: Oxymetazoline
- DENTAL - Full strength 0.5 mL (Experimental): Full strength oxymetazoline 0.5 mL to each naris (total = 500 mcg).
  Interventions: Drug: Oxymetazoline
- DENTAL - ½ strength 0.5 mL (Experimental): ½ strength oxymetazoline 0.5 mL to each naris (total = 250 mcg).
  Interventions: Drug: Oxymetazoline

INTERVENTIONS:
Drug: Oxymetazoline
  Other Names: Afrin

SUMMARY:
Oxymetazoline is an α-adrenergic agonist that is commonly used as a topical sympathomimetic agent in over-the-counter decongestant sprays. It is used extensively at Nationwide Children's Hospital for surgical procedures to produce vasoconstriction and reduce bleeding. Although there is generally limited vascular absorption, when administered in larger doses, uptake of oxymetazoline can lead to significant systemic hemodynamic effects. The NCH anesthesia department recently reported a case of oxymetazoline induced postoperative hypertension in a three-year-old child following inferior turbinate reduction and adenoidectomy. Current practice at NCH is to soak pledgets with full strength oxymetazoline and insert a varying number of pledgets during surgical procedures or instill oxymetazoline drops into the nose prior to nasotracheal intubation. There is no pediatric data regarding the method of administration and the absorption of oxymetazoline or the dose-response relationship of oxymetazoline serum levels on blood pressure and heart rate. These studies would be the first to determine safe and appropriate doses of oxymetazoline in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 2 through 12 yrs.
* Scheduled for: operative dentistry, functional endoscopic sinus surgery, or turbinate reduction (with or without tonsillectomy and/or adenoidectomy).

Exclusion Criteria:

* Treatment with oral decongestants or antihistamines within 24 hours of surgery.
* Taking anticoagulants.
* History of nasal trauma.
* History of epistaxis (nose bleeds).
* History of hypertension or cardiac disease.
* Allergy to oxymetazoline.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Oxymetazoline plasma concentration | 5, 10, 20, 45, 90 & 150 mins. after dosing

SECONDARY OUTCOMES:
Heart rate | Every 2-5 mins. for a maximum of 240 mins.
  Assessing for bradycardia
Blood pressure | Every 2-5 mins. for a maximum of 240 mins.
  Assessing for hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cartabuke, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States